CLINICAL TRIAL: NCT04798495
Title: Return to Everyday Life After Non-myeloablative Allogeneic Haematopoietic Stem Cell Transplantation; Feasibility and Participants' Perspectives of a Targeted Multimodal Interdisciplinary Rehabilitation Programme (HAPPY)
Brief Title: Feasibility of a Rehabilitation Programme Targeted Patients Treated With Non-myeloablative Stem Cell Transplantation
Acronym: HAPPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HAPPY-1
Record Dates: First submitted 2021-02-23; First posted 2021-03-15 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2020-12

CONDITIONS: Stem Cell Transplantation; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAPPY (Experimental): Single arm longitudinal design.
  Interventions: Other: Multimodal interdisciplinary rehabilitation programme (HAPPY)

INTERVENTIONS:
Other: Multimodal interdisciplinary rehabilitation programme (HAPPY) — A 6-month multimodal interdisciplinary rehabilitation programme abbreviated HAPPY was tested. The programme consisted of motivating interviewing technique, individual dialogues with fixed subjects, individual supervised physical exercise training, relaxation exercises, nutritional counselling, and group sessions (a combination of topics and exchange of experiences) with patients and relatives. To reach patients at home, the team phoned patients, who were also given tablets with access to the project's homepage and a digital physical exercise programme.

SUMMARY:
Non-myeloablative allogeneic haematopoietic stem cell transplantation (NMA-HSCT) is associated with innumerable complications and side-effects and a high treatment-related mortality. Maintaining quality of life, physical and psychosocial functioning and participation in society is therefore challenging for patients undergoing treatment with NMA-HSCT. This situation creates an urgent need for rehabilitation for patients to return to a meaningful everyday life, and for knowledge about how to best help this group of patients return to everyday life.

The project aims to develop and examine the feasibility and safety of a multimodal interdisciplinary rehabilitation programme targeted patients undergoing treatment with NMA-HSCT.

Three studies are planned. Study I is a qualitative interview study to get a profound insight into patients' experiences and challenges after NMA-HSCT.

Study II has a single arm longitudinal design with both a feasibility and an outcome component. Patients (N=30) are consecutively recruited at the Department of Haematology, Aarhus University Hospital, Denmark and enrolled in the 6-month HAPPY programme as soon as the decision about NMA-HSCT is final. Data is collected pre-NMA-HSCT, at 3-month, 6-month and 12-month after NMA-HSCT.

Study III is a qualitative interview study, where patients who participated in the rehabilitation programme evaluate the programme's influence on their return to everyday life.

The project contributes with knowledge about the feasibility of a rehabilitation programme targeted at a vulnerable group of chronic cancer patients with rare diseases. We will document the impact of an interdisciplinary intervention anchored in the hospital setting but aimed at reaching patients at home. If the intervention enhances quality of life, patient activation and functioning, it may not only reduce the number of hospitalizations and use of healthcare services, but may also allow more patients to maintain contact with the labour market and resume participation in society.

DETAILED DESCRIPTION:
Rehabilitation is becoming increasingly important in the face of growing diversity and intensity of cancer treatment and so is treatment with haematopoietic stem cell transplantation from a donor. Non-myeloablative allogeneic haematopoietic stem cell transplantation (NMA-HSCT) is associated with innumerable complications and side-effects and a high treatment-related mortality. Maintaining quality of life, physical and psychosocial functioning, and participation in society is therefore challenging for patients undergoing treatment with NMA-HSCT. This situation creates an urgent need for rehabilitation for patients to return to a meaningful everyday life, and for knowledge about how to best support this group of patients' return to everyday life.

The overall aim is to develop and evaluate the feasibility of a targeted multimodal interdisciplinary rehabilitation programme by involving patients undergoing NMA-HSCT.

Three studies were planned in accordance with the theoretical framework of Complex Interventions.

Study I is a qualitative focus group interview study using the Interpretive Description methodology. The purpose was to explore the experiences and perspectives of NMA-HSCT patients regarding their challenges and needs during their return to everyday life after HSCT transplantation.

Study II has a single arm longitudinal design with both a feasibility component and an outcome component.

The aim was to develop and to assess feasibility of the multimodal interdisciplinary rehabilitation programme HAPPY in patients with haematological cancers undergoing NMA-HSCT. Furthermore, to report health related quality of life, Patient Activation Measurement, cardiorespiratory capacity (VO2peak), muscle extension power, lean body mass, days at hospital, return to work and survival. A 6-month multimodal interdisciplinary rehabilitation programme was tested. The programme consisted of motivating interviewing technique, individual supervised physical exercise training, relaxation exercises, nutritional counselling, and group sessions (a combination of topics and exchange of experiences) with patients and relatives. To reach patients at home, the team phoned patients, who were also given tablets with access to the project's homepage and a digital physical exercise programme. Feasibility parameters were acceptability, exposure, fidelity, practicality, safety

Study III is a qualitative interview study using the Interpretive Description methodology. The aim was to explore patients' experiences and perspectives on relevance and meaning of participating in the multimodal interdisciplinary rehabilitation programme HAPPY, and the programme's influence on handling everyday life, during and after NMA-HSCT.

The project contributes with knowledge about the feasibility of a rehabilitation programme targeted at a vulnerable group of chronic cancer patients with rare diseases. We will document the impact of an interdisciplinary intervention anchored in the hospital setting but aimed at reaching patients at home. If the intervention enhances health related quality of life, patient activation and functioning, it may not only reduce the number of hospitalizations and use of healthcare services, but may also allow more patients to maintain contact with the labour market and resume participation in society.

ELIGIBILITY:
Inclusion Criteria:

* Patients were accepted for NMA-HSCT
* ≥ 18 years
* able to read and understand Danish and to follow the study protocol.

Exclusion Criteria:

* psychological diagnosis
* contra-indications for progressive exercise training
* inability to walk or stand
* instable bone lesions
* severe neurological deficiencies
* severe cardiac or cardio vascular diseases, severe pulmonary global insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Baseline - 6-month follow-up
  Number of patients who accepted to participate in the study out of patients treated with non-myeloablative allogeneic haematopoietic stem cell transplantation
Attrition and reasons for drop out | Baseline - 6-month follow-up
  Number of drop-outs of patients participating in the study
Exposure to physical exercise training per patient | Baseline - 6-month follow-up
  The percentage of physical exercise training used by the patients when he/she was at the hospital and reason(s) for non-participation
Exposure to motivating interviewing per patient | Baseline - 6-month follow-up
  The percentage of motivating interviewing used by the patients out all planned, and reason(s) for non-participation
Exposure to group sessions topics together with fellow patients and relatives per patient | Baseline - 6-month follow-up
  The percentage of group sessions with different topics used by the patients out all planned, and reason(s) for non-participation
Exposure to nutritional counselling per patient | Baseline - 6-month follow-up
  The percentage of nutritional counselling used by the patients out of planned, and reason(s) for non-participation
Exposure to digital physical exercise programme per patient | Baseline - 6-month follow-up
  The percentage usage of the digital exercise programme out of possible/planned digital exercise trainings, and reason(s) for non-participation
Exposure to phone calls to patients staying at home | Baseline - 6-month follow-up
  The percentage use of phone calls by patients while they stay at home, and reason(s) for unused
Exposure to individual dialogues | Baseline - 6-month follow-up
  The percentage of individual dialogues with fixed subjects used by the patients out all planned, and reason(s) for non-participation
Adverse Events | Baseline-1-year follow-up
  The number of adverse events related to the intervention

SECONDARY OUTCOMES:
Fidelity of physical exercise training | Baseline - 6-month follow-up
  The percentage of physical exercise trainings delivered as planned, and reason(s) for cancellation
Fidelity of motivating interviewing | Baseline - 6-month follow-up
  The percentage of motivating interviewing delivered as planned, and reason(s) for cancellation
Fidelity of individual dialogues | Baseline - 6-month follow-up
  The percentage of individual dialogues with fixed subjects delivered as planned, and reason(s) for cancellation
Fidelity of group sessions | Baseline - 6-month follow-up
  The percentage of group sessions with different topics and exchange of experiences delivered as planned, and reason(s) for cancellation
Fidelity of nutritional counselling | Baseline - 6-month follow-up
  The percentage of nutritional counselling delivered out of planned, and reason(s) for cancellation
Fidelity of the digital exercise programme | Baseline - 6-month follow-up
  The percentage delivery of the digital exercise programme out of planned digital exercise trainings, and reason(s) for cancellation
Fidelity of delivered phone calls | Baseline - 6-month follow-up
  The percentage of delivered phone calls to patients at home, , and reason(s) for cancellation
Practicability of questionnaires and physical tests | Baseline-1-year follow-up
  Percentage of questionnaires and physical tests performed out of possible questionnaires and physical tests, and reason(s) for delay or cancellation

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Lindman, Principal Investigator — Aarhus University Hospital
Locations (1):
- Dep. of Hem. Aarhus Universitetshospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No